CLINICAL TRIAL: NCT05582473
Title: Pilot Test of Juntos/Together Program to Build Confidence for Complex Care Tasks Among Latino Family Caregivers
Brief Title: Juntos/Together Program to Build Confidence for Complex Care Tasks Among Latino Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC20220579H
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Dementia Caregivers
Keywords: Latino caregivers

STUDY DESIGN:
Intervention Model Description: A randomized wait-list control group design with blinded outcomes assessment to examine the effectiveness of LST-LC on caregiver confidence and self-efficacy in performing complex care tasks. This design has the advantage of making enrollment more feasible as participants may find the intervention highly desirable and will eventually receive it. Yet, the design provides a randomized comparison with a non-intervention control group. Participants will be individually randomized 1:1 to an immediate intervention group (IG) and a wait-list (delayed) control group (WLC).
Who Masked: Outcomes Assessor
Masking Description: The research assistant will collect follow-up data and will be blinded to group assignment. Caregivers will be asked not to discuss whether they were in a group program prior to follow-up data collection with the research assistant. The statistician will also be blinded, with group assignment designated using a binary variable in anonymous study data. In order to conduct study activities, other team members will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-List Control Group (No Intervention): Randomized subjects will wait for a 3 month period before being assigned to the LST-LC education. This group of subjects will act as the control group.
- Learning Skills Together-Latino Caregivers (LST-LC) (Other): The study team convened a team of health care professionals, including nursing, occupational therapy, speech-language pathology, gerontology, nutrition, and dental hygiene, to develop a community-based education program for family caregivers.
  Interventions: Behavioral: LST-LC Education

INTERVENTIONS:
Behavioral: LST-LC Education — Testing the LST-LC intervention with cultural adaptations integrated through Stage 2 (Adaptation Design). There are 9 modules.
  Session 1, we describe the principles underlying the program (safety, hygiene, dignity, comfort, and independence), discuss self-care, and introduce a vignette of caring for a person with dementia, designed to generate conversation around the caregiving role.
  Other modules focus on 1) behavioral and 2) communication challenges in the context of dementia; 3) home safety, transfers, and adaptable medical equipment; 4) managing nutrition needs; 5) swallowing challenges; 6) supporting oral hygiene; 7) dealing with incontinence, including preventing and recognizing urinary tract infections; 8) medication management and 9) managing comorbidities including assessing and managing pain
  Arms: Learning Skills Together-Latino Caregivers (LST-LC)

SUMMARY:
The overall goal of this study is to culturally adapt and test the effectiveness of Learning Skills Together (LST) in improving self-efficacy among Latino family caregivers. To address this overall goal, the study team propose the following aims: i) culturally adapt the LST intervention for Latino caregivers using a community-engaged approach; and ii) examine the effect of the LST intervention on Latino caregiver self-efficacy, depression, and well-being using a randomized wait-list control group.

DETAILED DESCRIPTION:
The study team will use a randomized wait-list control group design with blinded outcomes assessment to examine the effectiveness of LST-LC on caregiver confidence and self-efficacy in performing complex care tasks. This design has the advantage of making enrollment more feasible as participants may find the intervention highly desirable and will eventually receive it. Yet, the design provides a randomized comparison with a non-intervention control group. Participants will be individually randomized 1:1 to an immediate intervention group (IG) and a wait-list (delayed) control group (WLC).

ELIGIBILITY:
Inclusion Criteria:

1. a family member to an individual living with AD/ADRD (Alzheimers Disease/Alzheimers Disease and related dementias) who has received a diagnosis from a physician,
2. aged 18 years or older,
3. providing assistance with at least two instrumental activities of daily living or one activity of daily living,
4. providing care to a person with dementia in mid-stage as defined by a score between 4 and 6 on the Global Deterioration Scale (GDS), and
5. not paid to provide care

Exclusion Criteria:

1. are unable to read and speak English or Spanish,
2. previously participated in LST, and/or
3. have plans to place the care recipient in a skilled nursing facility within the next 6 months (i.e., study duration).
4. Participants must have a Patient Health Questionnaire (PHQ-9) score of less than 15, the threshold for moderately severe depression
5. Participants with severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Self-Efficacy Scale | Baseline to 6 weeks
  This is a unidimensional measure, with total score ranging between 1 and 10, with mean (SD) of 6.0 (2.1) in a sample of 158 caregivers (Ritter et al., 2022). Higher scores indicate higher confidence.

SECONDARY OUTCOMES:
Complex Care Tasks Scale | Baseline to 6 weeks
  A scale developed by the study team with total score ranging from 14 to 70. Items are summed and averaged. In our pilot study with 35 caregivers, the mean (SD) was 3.7 (0.8) (Meyer et al., 2022). Higher scores indicate higher confidence.
Caregiver Confidence in Medical Sign/Symptom Management (CCSM) scale | Baseline to 6 weeks
  A 25 item scale which evaluates the efforts to support family caregivers of people with dementia in their daily medical management responsibilities requires a measure of caregiver self-efficacy (confidence).The total score on this scale ranges from 25 to 125, with items summed and averaged with a mean (SD) of 3.8 (0.6) in a sample of 194 caregivers (Zimmerman et al., 2018). Higher scores indicate higher confidence.

OTHER OUTCOMES:
Patient Reported Outcomes Measurement Information systems (PROMIS) Global Health Score | Baseline to 6 weeks
  For this scale, each of the each of the individual 10 items can be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health, and general perceptions of health (ranging from 1 to 5) with higher scores indicating better global health. There are also two-subscales, Physical Health (PH) and Mental Health (MH) that can be converted to standardized T-score values, with a T-score of 50 which represents the mean of the general population and higher scores indicate better physical and mental health.
Lubben Social Network Scale (LSNS-6) | Baseline to 6 weeks
  A six item, self reported scale to assess social isolation in older adults by measureing perceived social support received by family and friends. The total score is calculated by finding the sum of the all items, with the score ranges between 0 and 30, with a higher score indicating more social engagement.
Revised Memory and Behavior Checklist | Baseline to 6 weeks
  A 24-item scale used to measure behavioral challenges experienced by the person living with dementia, from the perspective of the caregiver. The possible range for this scale is 0-96, the mean frequency (SD) of behaviors is 34 (16.6) and the mean reaction (SD) is 22.7 (15.6). A lower score indicates better coping skills.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L White, PhD, BSN, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The community-engaged approach used to adapt and test the intervention will also support dissemination. The investigators will work closely with community-based organizations such as the local Area Agency on Aging and Alzheimer's Association for recruitment and , will provide quarterly updates to community partners on progress through the Family Caregiver Coalition and Caring for the Caregiver newsletters. The investigators will disseminate the results of the study through community forums, as well as publication in peer-reviewed journals and presentations at professional meetings. The target audience for dissemination is community organizations who support family caregivers. With that in mind, we will target the American Society on Aging for presenting the results of the study.
  Information will be shared as a publication in a peer reviewed scientific journal
Supporting Information: Study Protocol, SAP
Time Frame: After data collected during the study has been analyzed and published.